CLINICAL TRIAL: NCT03655665
Title: Does the Use of Topical Otic Drops at the Time of Tympanostomy Tube Placement Improve Outcomes When no Middle Ear Effusion is Present at the Time of Surgery
Brief Title: Does Topical Otic Drop Use at Time of Tympanostomy Tube Surgery Improve Outcomes When no Middle Ear Effusion is Present
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Kenneth Whittemore, Associate Otolaryngologist/Assistant Professor of Otolaryngology, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P00026372
Record Dates: First submitted 2018-08-22; First posted 2018-08-31 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Otitis Media
MeSH Terms: conditions — Otitis Media | interventions — Ofloxacin

STUDY DESIGN:
Intervention Model Description: Clinical effectiveness model. Each subject will serve as their own control. Subject's ears will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Ear (Experimental): Participants will serve their own control. Participants will receive 3 drops of ofloxacin otic solution intra- and post-operatively 3 times per day for 3 days in ONE ear. Ear sidedness will be randomized by participant.
  Interventions: Drug: Ofloxacin otic solution
- No Intervention (No Intervention): Participants will serve their own control. Participants will receive no intervention in the ear contralateral to the treated ear. Ear sidedness will be randomized by participant.

INTERVENTIONS:
Drug: Ofloxacin otic solution — Three drops of ofloxacin otic 0.3%. intra and post-operatively for 3 days post-surgery on one ear.
  Other Names: Floxin Otic
  Arms: Treatment Ear

SUMMARY:
To determine whether the use of topical otic drops intra-operative and post-operative during tympanostomy tube placement reduces the rate of tympanostomy tube occlusion and post-operative otorrhea (ear drainage) during the initial 4-week post-operative period in subjects with no middle ear effusion (fluid behind the ear drum) present at the time of surgery. A within subject controlled study design will be utilized to study this effect. Subjects with absent middle ear effusion who are receiving tympanostomy tube placement will receive a standard protocol of Floxin topical drops during surgery and after surgery in one ear. Selection of ear (right ear or left ear) will be randomized. The primary measured outcome will be the rate of tympanostomy tube occlusion within first 4 weeks postoperatively. The secondary measured outcome is the rate of tympanostomy tube otorrhea (drainage) within first 4 weeks postoperatively.

DETAILED DESCRIPTION:
Background and Significance: Two major factors affecting the delivery of quality patient care today are cost of care and development of antibiotic resistance. If no significant difference is found in the rate of tympanostomy tube occlusion and drainage in subects receiving ear drops after surgery and those not receiving ear drops, may help prevent the development of antibiotic resistance and could possibly reduce the cost of care for families.

Tympanostomy tube(s) (TT) insertion is the most common otolaryngologic procedure for children and adolescents who suffer from chronic otitis media. TT(s) are inserted by a surgeon through the eardrum to regulate pressure in the middle ear and to aid with ear drainage and ventilation. In order for TT(s) to ventilate the middle ear space properly, they must remain unobstructed. Otorrhea is one of the most common complications following TT(s) insertion. Previous research has suggested that various factors may lead to TT(s) occlusion, including blood, debris, purulent otorrhea and tube size. A 2014 study by Conrad et al., found that patients with the presence of middle ear effusion at the time of surgery were more likely to experience tube occlusions than patients without fluid. However, studies demonstrating the most effective treatment for preventing postoperative otorrhea and TT occlusion are limited.

How to reduce the risk of post-operative TT otorrhea and TT occlusion is a common question among otolaryngologists and researchers and the efficacy of ototopical drops has been debated for patients without middle ear fluid. There is conflicting information in the current literature about the utility of these topical otic drops in patients with dry ears on the day of surgery. A 2008 review of seven randomized controlled trials completed by Schmelzle and colleagues concluded that fluoroquinolone based topical otic drops are the most effective treatment for patients with acute otitis media and TTs when compared to systemic antibiotic treatment and placebo. However, this treatment has been long debated. A 1991 study published by Ramadan, Tarazi, and Zaytoun found that there was no statistical difference between treated vs. not treated group in the development of post-operative otorrhea; however, all of these patients had middle ear effusions at the time of TT placement. Concurrently, a 2009 ex vivo study by Burke and colleagues on clotted TT(s) found that the administration of a solution of vinegar and hydrogen peroxide produced patent tubes at a higher rate than antibiotic otic drops.

Additionally, antibiotic resistance is a growing concern when treating with oral antibiotic therapy. While the placement of tympanostomy tubes does reduce the need for oral antibiotic therapy, resistant strains of bacteria such as methicillin-resistance staphylococcus aureus (MRSA) have become more prevalent in children with tympanostomy tubes.

Given the lack of evidence-based research, the decision for usage of topical otic drops when there is no middle ear fluid present is based on the subject's medical history and clinical judgment of the treating physician. Some providers opt to use topical otic drops in the absence of middle ear effusion, and some providers forgo the use of drops intra- and/or post-operatively. When topical otic drops are used as part of standard of care they are placed bilaterally, and patients receive variable amounts of otic solution intra- and post-operatively, also based on clinician preference.

Some providers believe that the use of topical otic drops in the absence of middle ear fluid effectively lessens the potential of a post-operative negative outcome such as TT occlusion. If this is true, not using topical otic drops intra- or post-operatively exposes the patient to a higher risk of a negative surgical outcome. However, there is currently insufficient clinical evidence to support the efficacy of topical drops in that specific clinical scenario. If indeed topical otic drops do not effectively improve post-operative outcomes, then the use of them is exposing the patient to antibiotics and adding to the cost of their care unnecessarily. The goal of this present study is to demonstrate whether the use of topical ofloxacin otic drops in patients with absent middle ear effusion on the day of TT surgery impacts the development of post-operative tube otorrhea or occlusion.

In the proposed study, subjects' ears will be randomized and ofloxacin drops will be administered intra- and post-operatively in either their left or right ear, depending on treatment group. Subjects will be followed-up at their 4-week appointment to determine presence of otorrhea and patency of tubes.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a history of Eustachian tube dysfunction (ETD) or recurrent acute otitis media (AOM) requiring surgery for bilateral TT placement
* Participant's caregiver understands the protocol and is willing to comply with the protocol
* Children ages 6 months to 10 years undergoing surgery for bilateral tympanostomy tube placement without middle ear fluid on the day of their surgery

Exclusion Criteria:

* Participant is having concomitant procedures performed at the time of their tympanostomy tube surgery (i.ei.e. adenoidectomy, airway endoscopy, nasal cautery).
* Historyof conductive hearing loss, as determined from their last audiogram prior to tympanostomy tube procedure
* Middle ear effusion present in either their left or right ear on the day of tympanostomy tube surgery
* Current diagnosis of craniofacial abnormalities, Trisomy 21, primary ciliary dyskinesia, cystic fibrosis
* History of a known immunodeficiency disease

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with tympanostomy tube occlusion | 0-35 days post-op
  Any non-"large volume" ear canal volume (less than 1.00cc volume) measurement at 4 week visit, in conjunction with physical examination notable for occluded TT, would be consistent with tube occlusion.

SECONDARY OUTCOMES:
Percentage of patients with otorrhea (drainage from the ear) | 0-35 days post-op
  Any drainage of liquid from the ear. Can be clear, bloody, or purulent

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R. Whittemore, MD, MS, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital at Waltham, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenfeld RM, Schwartz SR, Pynnonen MA, Tunkel DE, Hussey HM, Fichera JS, Grimes AM, Hackell JM, Harrison MF, Haskell H, Haynes DS, Kim TW, Lafreniere DC, LeBlanc K, Mackey WL, Netterville JL, Pipan ME, Raol NP, Schellhase KG. Clinical practice guideline: Tympanostomy tubes in children. Otolaryngol Head Neck Surg. 2013 Jul;149(1 Suppl):S1-35. doi: 10.1177/0194599813487302. PMID 23818543
- [Background] Kay DJ, Nelson M, Rosenfeld RM. Meta-analysis of tympanostomy tube sequelae. Otolaryngol Head Neck Surg. 2001 Apr;124(4):374-80. doi: 10.1067/mhn.2001.113941. PMID 11283489
- [Background] van Dongen TM, van der Heijden GJ, Freling HG, Venekamp RP, Schilder AG. Parent-reported otorrhea in children with tympanostomy tubes: incidence and predictors. PLoS One. 2013 Jul 12;8(7):e69062. doi: 10.1371/journal.pone.0069062. Print 2013. PMID 23874870
- [Background] Jeon EJ, Park YS, Lee SK, Chang KH, Park SY, Park KH, Lee DH. Factors of the blockage of ventilation tubes in the immediate postoperative period. Eur Arch Otorhinolaryngol. 2007 Dec;264(12):1393-7. doi: 10.1007/s00405-007-0375-0. Epub 2007 Jul 27. PMID 17657506
- [Background] Jamal TS. Avoidance of postoperative blockage of ventilation tubes. Laryngoscope. 1995 Aug;105(8 Pt 1):833-4. doi: 10.1288/00005537-199508000-00012. PMID 7543180
- [Background] Schmelzle J, Birtwhistle RV, Tan AK. Acute otitis media in children with tympanostomy tubes. Can Fam Physician. 2008 Aug;54(8):1123-7. PMID 18697973
- [Background] Conrad DE, Levi JR, Theroux ZA, Inverso Y, Shah UK. Risk factors associated with postoperative tympanostomy tube obstruction. JAMA Otolaryngol Head Neck Surg. 2014 Aug;140(8):727-30. doi: 10.1001/jamaoto.2014.1176. PMID 25009981
- [Background] Ramadan HH, Tarazi T, Zaytoun GM. Use of prophylactic otic drops after tympanostomy tube insertion. Arch Otolaryngol Head Neck Surg. 1991 May;117(5):537. doi: 10.1001/archotol.1991.01870170083018. PMID 2021473
- [Background] Burke EL, Walvekar RR, Lin J, Hagan J, Kluka EA. Common agents used to unblock blood clots within tympanostomy tubes: an ex vivo study and review of literature. Int J Pediatr Otorhinolaryngol. 2009 Dec;73(12):1725-8. doi: 10.1016/j.ijporl.2009.09.009. Epub 2009 Sep 30. PMID 19796828
- [Background] Giles W, Dohar J, Iverson K, Cockrum P, Hill F, Hill N. Ciprofloxacin/dexamethasone drops decrease the incidence of physician and patient outcomes of otorrhea after tube placement. Int J Pediatr Otorhinolaryngol. 2007 May;71(5):747-56. doi: 10.1016/j.ijporl.2007.01.012. Epub 2007 Feb 20. PMID 17316832